CLINICAL TRIAL: NCT03844633
Title: Initiation of Injectable Contraception Immediately Postpartum Among Breastfeeding Women
Brief Title: Postpartum Family Planning
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Because of insufficient enrollment, we closed the RCT and replaced it with an observational design
Sponsor: Ohio State University (Other)
Collaborators: Nationwide Children's Hospital (Other); Emory University (Other)
Responsible Party: Principal Investigator, Maria F. Gallo, PhD, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017H0445
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Delay in Time to Lactogenesis Stage II
Keywords: lactation; Depo Provera; contraception
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The intervention and control injection arms will be blinded. The no injection arm will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Intervention arm (Experimental): Intramuscular injectable depot medroxyprogesterone acetate (1 mL of medroxyprogesterone acetate sterile aqueous suspension 150 mg/mL) provided within 48 hours of childbirth
  Interventions: Drug: Depo-Provera Injectable Product
- Placebo arm (Placebo Comparator): 0.9% sodium chloride injection provided within 48 hours of childbirth
  Interventions: Drug: Placebos
- Open arm (No Intervention): No intervention provided

INTERVENTIONS:
Drug: Depo-Provera Injectable Product — Depo-Provera Injectable Product -- Shot administered within 48 hours of childbirth
  Arms: Intervention arm
Drug: Placebos — Placebos -- Shot administered within 48 hours of childbirth
  Arms: Placebo arm

SUMMARY:
Investigators will conduct a randomized controlled trial (RCT) to evaluate the effects of immediate postpartum initiation of DMPA on breastfeeding and long-term contraceptive use. Investigators will randomize approximately 429 adult women who have delivered a healthy, full-term infant at The Ohio State University Wexner Medical Center (OSUWMC), who intend to breastfeed for ≥6 months, and who want to use DMPA (Depo-Provera; Pfizer Corp.) Note that because of anticipated screening failures, investigators will enroll more than the number randomized (i.e., up to 800 women). Investigators will randomize women to receive within 48 hours of delivery: 1) DMPA ("intervention" arm), 2) placebo injection ("placebo" arm) or 3) no injection ("open control" arm). The first two arms will be blinded while the open control arm will be unblinded. Note that postpartum patients at the study site do not receive DMPA before discharge as standard care. At enrollment, women will receive condom counseling and provision and referral for contraception at 12 weeks (intervention and placebo arms) or at 6 weeks postpartum (open control arm). Investigators will collect data on lactogenesis, infant feeding and growth, and contraception use during 12 follow-up months. Investigators conducted a pilot study (N=100) in the target population, which supports the feasibility of the current trial.

DETAILED DESCRIPTION:
Postpartum women often are inadequately protected against rapid repeat pregnancy. Ensuring adequate inter- birth intervals could prevent an estimated 9% of deaths worldwide among children less than 5 years of age. Intramuscular injectable depot medroxyprogesterone acetate (DMPA) is rapidly becoming the method of choice in some settings, including regions where high maternal and child mortality make birth spacing critical. DMPA possesses many advantages for postpartum contraception as compared to other methods. However, the World Health Organization (WHO) advises against use of progestin-only injectables during the first six weeks postpartum among breastfeeding women. In contrast, the Centers for Disease Control and Prevention (CDC) recommends that progestin-only injectables generally can be started immediately postpartum on the grounds that their known advantages, as a whole, outweigh their unknown risks. This inconsistency in guidance reflects the lack of high-quality data for making evidence-based decisions. Studies conducted, to date, have important limitations: short follow-up intervals, low power, lack of consistency in using sensitive and standardized assessments, and lack of randomized trials evaluating DMPA administration specifically in the immediate postpartum period. Investigators propose to evaluate the effects of immediate postpartum initiation of DMPA on breastfeeding and on child development. We will conduct a randomized controlled trial of 429 adult women who have delivered a healthy, full-term infant, intend to breastfeed for ≥6 months, and want to use DMPA. Women will be randomized to receive within 48 hours of delivery: 1) DMPA ("intervention" arm), 2) placebo injection ("placebo" arm) or 3) no injection ("open control" arm). The first two arms will be blinded while the open control arm will be unblinded. Investigators will determine the effect of immediate postpartum initiation of DMPA on breastfeeding (Aim 1) and on contraception use (Aim 2). The proposed trial is innovative in use of 1) a randomized, partially-blinded design with sufficient power and follow up; 2) standardized, validated measures on lactation as well as breastfeeding and contraception behaviors; and 3) whole-body air displacement plethysmography to identify differences between arms in infant body composition. The findings of a pilot study in the target population support the feasibility of the proposed trial. Investigators expect the trial findings will permit the harmonization of the WHO and CDC guidance on the timing of DMPA initiation among breastfeeding women. This would have important implications for shaping global policy and practice worldwide, especially in settings where inadequate birth spacing contributes to high maternal and infant morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Intend to deliver in the Labor and Delivery Unit at Ohio State University Wexner Medical Center, Grady Memorial Hospital or Emory University Midtown;
2. Are ≥18 years of age;
3. Speak English;
4. Intend to breastfeed, or express milk for their infant, for ≥6 months;
5. Do not want to become pregnant within the first 12 months after delivery;
6. Want to start use of DMPA immediately after delivery before discharge or no hormonal contraception immediately postpartum; AND
7. Intend to reside in Ohio or Georgia for the first 12 months after delivery.

   Exclusion Criteria:
8. Undiagnosed vaginal bleeding;
9. Known or suspected malignancy of breast;
10. Active thrombophlebitis, or current or past history of thromboembolic disorders, or cerebral vascular disease;
11. Liver dysfunction or disease; OR
12. Known hypersensitivity to Depo-Provera.

Women who enroll prenatally will need to rescreen following delivery to confirm their eligibility. Women enrolling after delivery or who are rescreening will need to meet criteria 2-12 above as well as the following eligibility criteria:

1. Are a postpartum patient in the Labor and Delivery Unit at OSUWMC, Grady Memorial Hospital or Emory University Midtown Hospital; AND
2. Have delivered a term, singleton infant of ≥2500 grams without any apparent health concerns.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2022-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gallo, PhD, Principal Investigator — The Ohio State University, College of Public Health
Locations (1):
- Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
We will welcome collaboration with others who could make use of the study materials and study datasets resulting from the project. Once the primary results are accepted for publication in a peer-reviewed journal, we will make full, de-identified datasets available to individual investigators formally requesting this access.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Once the primary results are accepted for publication in a peer-reviewed journal, we will make full, de-identified datasets available to individual investigators formally requesting this access.
Access Criteria: The request should specify the data variables needed, the plan for their analysis, the individuals who will have access to the data, and the plan for destroying the data once the planned analysis is completed. To protect the integrity of the data, the requestor must submit proof of IRB approval or exemption from their institution before we will release the data. The shared data will not contain any individual participant identifiers. The data will be sent in a secured encrypted data file, and the requestors will be responsible for notifying the project PIs upon completion of analysis and specifying the manner in which the data were destroyed. Any presentations, abstracts, or publications will be required to include an acknowledgement of the trial funding source.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 enrolled participant was missing data on their assigned arm.
Period: 1 Week FU
Arm/Group | Intervention Arm | Placebo Arm | Open Arm
Started | 16 | 15 | 17
Completed | 16 | 14 | 13
Not Completed | 0 | 1 | 4
Not completed — Lost to Follow-up | 0 | 1 | 4
Period: 12-month Follow-up
Arm/Group | Intervention Arm | Placebo Arm | Open Arm
Started | 16 | 15 | 17
Completed | 9 | 10 | 9
Not Completed | 7 | 5 | 8
Not completed — Lost to Follow-up | 7 | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Placebo Arm | Open Arm | Total
Number analyzed (Participants) | 16 | 15 | 17 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.9 (4.5) | 29.3 (5.9) | 29.1 (5.1) | 29.1 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 17 | 48
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 16 | 13 | 16 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 8 | 10 | 24
  White | 8 | 6 | 7 | 21
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 15 | 17 | 48
Study site [Count of Participants; unit: Participants]
  Columbus, OH | 14 | 14 | 14 | 42
  Atlanta, GA | 2 | 1 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Time to Lactogenesis Stage 2
Description: Self-reported time to lactogenesis stage 2 (i.e., milk "let-down")
Time Frame: within 7 days postpartum
Measure: Mean (Full Range); unit: hours
Arm/Group | Intervention Arm | Placebo Arm | Open Arm
Number analyzed (Participants) | 16 | 14 | 13
hours | 44.8 [11.3 to 125.6] | 47.2 [1.5 to 112.0] | 50.4 [1.0 to 103.4]

2. Primary Outcome: Use of Highly-effective Contraception
Description: Rates of use of a highly-effective method of contraception (defined here as DMPA, implant, IUD, sterilization, pill, patch, or ring) at 12 months post-delivery among women in the intervention or placebo arm versus those in the open control arm
Time Frame: At 12 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm | Open Arm
Number analyzed (Participants) | 9 | 10 | 9
Participants | 7 | 6 | 4

ADVERSE EVENTS:
Time Frame: One year from enrollment
Arm/Group | Intervention Arm | Placebo Arm | Open Arm
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT03844633/Prot_SAP_ICF_001.pdf